CLINICAL TRIAL: NCT01404650
Title: A Phase II Study of Hsp90 Inhibitor AUY922 for the Treatment of Patients With Refractory Gastrointestinal Stromal Tumor
Brief Title: Study of Hsp90 Inhibitor AUY922 for the Treatment of Patients With Refractory Gastrointestinal Stromal Tumor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI GI 148
Record Dates: First submitted 2011-07-21; First posted 2011-07-28 (Estimated); Results first posted 2016-10-04 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-08

CONDITIONS: Gastrointestinal Stromal Tumor
Keywords: GIST; Refractory; Gastrointestinal; Stromal; Tumor
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Neoplasms | interventions — 5-(2,4-dihydroxy-5-isopropylphenyl)-4-(4-morpholin-4-ylmethylphenyl)isoxazole-3-carboxylic acid ethylamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AUY922 (Experimental)
  Interventions: Drug: AUY922

INTERVENTIONS:
Drug: AUY922 — AUY922: 70 mg/m2 IV over 60 minutes on Days 1, 8, and 15 of each cycle. Treatment cycles will be repeated every 21 days. Patients will be evaluated for response at 6 and 12 weeks and then every 9 weeks (i.e., every 3 cycles) thereafter. Patients may continue treatment until evidence of disease progression.

SUMMARY:
This is a multicenter, non-randomized, single agent, Phase II study of AUY922 in patients with refractory Gastrointestinal Stromal Tumor (GIST). The primary endpoint of this study is to determine progression-free survival (PFS) for patients with GIST receiving AUY922 intravenously (IV) on Days 1, 8, and 15 of a 21-day treatment cycle with restaging at 6 and 12 weeks and then every 9 weeks thereafter. Patients may continue treatment until evidence of disease progression.

DETAILED DESCRIPTION:
Gastrointestinal stromal tumors (GIST) are common sarcomas that arise in the gastrointestinal tract. Sunitinib (Pfizer) and imatinib (Novartis) are FDA-approved for treatment of patients with GIST. However, patients with advanced or refractory GIST who are resistant to these agents eventually experience disease progression or death. Heat shock protein-90 (Hsp90) is a substance found in various malignancies that encourages tumor cells to grow and survive. As an inhibitor of Hsp90, AUY922 may decrease growth of tumor cells that were resistant to prior therapies. This study investigates AUY922 monotherapy as treatment for patients who either progressed on, or were resistant to, imatinib and sunitinib.

ELIGIBILITY:
Inclusion Criteria:

1. Pts with histologically-confirmed metastatic or unresectable GIST who have progressed on, are intolerant of, or are not a candidate for imatinib and sunitinib therapy. Pts must not have received prior treatment with Hsp90 inhibitors.
2. Must have an ECOG Performance Status of 0-1.
3. Must have a life expectancy of ≥3 mos.
4. Must have at least one unidimensional measurable lesion definable by MRI or CT scan. Disease must be measurable per RECIST v1.1.
5. Must have normal serum phosphorus and magnesium ≥ the lower limit of normal prior to trial entry.
6. Normal bone marrow function defined as: ANC ≥1500/μL Hgb ≥9 g/dL Plt ≥100,000/L
7. Adequate hepatic function defined as: AST or ALT and ALP must be 2.5 x ULN, or ≤5 x ULN in pts with liver mets Total bilirubin ≤1.5 x the institutional ULN
8. Renal function defined as: Serum creatinine ≤1.5 x ULN or 24-hour CrCl 50 mL/min
9. Women of childbearing potential (WOCP) must have a negative serum or urine pregnancy test performed ≤7 days prior to start of treatment.
10. Must be accessible for treatment and follow-up.
11. Must be able to understand the investigational nature of this study and give written informed consent prior to study entry

Exclusion Criteria:

1. Currently receiving or have received cancer therapies ≤21 days of initiating study therapy. For pts receiving small molecule targeted therapy, study treatment may begin ≥21 days after last dose or ≥5 half lives of previous treatment, whichever is shorter. The patient must have recovered from or come to a new chronic stable baseline from all treatment-related toxicities.
2. Use of any non-approved or investigational agent ≤30 days of administration of the first dose of study drug. Pts may not receive any other investigational or anti-cancer treatments while participating in this study.
3. Uncontrolled brain mets. Pts with treated brain mets (resection or radiotherapy) are eligible if brain mets have responded to treatment as documented by CT or MRI scan obtained at ≥2 wks after completion of RT, neurologic symptoms are absent, and steroids have been discontinued.
4. Treatment with therapeutic doses of coumadin-type anticoagulants (maximum daily dose of 1 mg allowed for port line patency permitted).
5. Impaired cardiac function with any one of the following: History (or family history) of prolong QT syndrome. Mean QTc ≥450 msec on baseline ECG. History of clinically manifested IHD ≤6 mos prior to study start. History of heart failure or any history of left ventricular (LV) dysfunction (LVEF ≤45%) by MUGA or ECHO. Clinically significant ECG abnormalities including 1 or more of the following: left bundle branch block, right bundle branch block with left anterior hemiblock. ST segment elevation or depression >1 mm, or 2nd (Mobitz II) or 3rd degree AV block. History or presence of A-Fib, atrial flutter or ventricular arrhythmias including ventricular tachycardia or Torsades de Pointes. Other clinically significant heart disease. Clinically significant resting bradycardia (<50 beats per minute). Currently receiving treatment with any medication which has a relative risk of prolonging the QTcF interval or inducing Torsades de Pointes and cannot be switched to an alternative drug or discontinued prior to commencing AUY922. Obligate use of a cardiac pacemaker.
6. Known diagnosis of HIV, Hep C virus, or acute or chronic Hep B infection.
7. Concurrent severe, intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements.
8. Women who are pregnant or lactating.
9. Any condition that would prevent patient comprehension of the nature of, and risk associated with, the study, and the inability to comply with study and/or follow-up procedures.
10. Other malignancies ≤3 years, with the exception of adequately treated basal or squamous cell carcinomas of the skin, carcinoma in situ of the cervix, or localized prostate cancer with a current PSA of <1.0 mg/dL on 2 successive evaluations, at least 3 mos apart, with the most recent evaluation no more than 4 wks prior to entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Bendell, MD, Study Chair — SCRI Development Innovations, LLC
Locations (8):
- United States (8):
  - Yale School of Medicine, New Haven, Connecticut
  - Florida Cancer Specialists-South, Fort Myers, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Woodlands Medical Center, Pensacola, Florida
  - Florida Cancer Specialists-North, St. Petersburg, Florida
  - Research Medical Center, Kansas City, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Tennessee Oncology, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multi-center trial evaluated AUY922 monotherapy as treatment for patients with gastrointestinal stromal tumor (GIST) refractory to, or intolerant of, imatinib and sunitinib. Between Dec 2011 and Jan 2015, 25 patients enrolled in the trial. Thirty-four patients (34) were planned to be enrolled but enrollment stopped early due to slow accrual.
Groups:
- AUY922: AUY922: 70 mg/m2 IV over 60 minutes on Days 1, 8, and 15 of each cycle. Treatment cycles repeated every 21 days. Patients are evaluated for response at 6 and 12 weeks and then every 9 weeks (i.e., every 3 cycles) thereafter until evidence of disease progression or intolerable toxicity.
Period: Overall Study
Arm/Group | AUY922
Started | 25 (Twenty-five patients received a median of 2 cycles of AUY922.)
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | AUY922
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 9
Age, Continuous [Median (Full Range); unit: years] | 63 [20 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Measured from time of randomization until objective tumor progression or death; assessed according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria. Progressive disease (PD) defined as at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest (nadir) sum since the treatment started, or the appearance of one or more new lesions.
Time Frame: At 6 and 12 weeks then every 9 weeks thereafter until progression or intolerable toxicity, up to 4 years.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AUY922
Number analyzed (Participants) | 25
months | 3.9 [2.5 to 5.3]

2. Secondary Outcome: Response Rate (RR)
Description: Defined as the proportion of complete and partial responses, assessed per RECIST v1.1. Complete response (CR) defined as a disappearance of all lesions; partial response (PR) defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking the baseline sum LD as reference. Stable Disease (SD) defined as neither sufficient shrinkage to qualify for PR, nor sufficient increase to qualify for progressive disease, taking as reference the smallest (nadir) sum LD since start of treatment.
Time Frame: At 6 and 12 weeks then every 9 weeks thereafter until progressive disease or intolerable toxicity, for up to 4 years.
Population: Of 25 patients enrolled, 4 patients were not evaluable for response due to treatment discontinuation prior to first disease evaluation.
Measure: Number; unit: percentage of participants
Arm/Group | AUY922
Number analyzed (Participants) | 21
percentage of participants
  Stable Disease | 60
  Objective Response | 4
  Progressive Disease | 20

3. Secondary Outcome: Overall Survival (OS)
Description: Evidence of survival was obtained by clinic visit or telephone contact from the time of first dose until death from any cause.
Time Frame: Every 3 months until patient death or lost to follow-up, for up to 4 years.
Population: All 25 patients who received treatment were included in the analysis of overall survival.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | AUY922
Number analyzed (Participants) | 25
months | 8.5 [5.2 to 16.7]

4. Secondary Outcome: Number of Patients With Adverse Events as a Measure of Safety and Tolerability
Description: Worst toxicity grades per patient were tabulated for select adverse events according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v 4.0
Time Frame: Days 1, 8 and 15 of each 21-day cycle plus 30 days after treatment discontinuation.
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | AUY922
Number analyzed (Participants) | 25
participants
  Anemia | 10
  Leukopenia | 1
  Thrombocytopenia | 1
  Diarrhea | 16
  Fatigue | 13
  Nausea | 11
  Vomiting | 7
  Asthenia | 5
  Abdominal Pain | 3
  Headache | 3
  Pain | 3
  Alkaline phosphatase increased | 2
  Anorexia | 2
  Dehydration | 2
  Dysgeusia | 2
  Blurred vision | 9
  Flashing lights | 7
  Delayed light/darl adaptation | 4
  Night Blindness | 3
  Floaters | 2
  Decreased color perception | 2
  Light sensitivity | 4
  Vision darkening | 2
  Vision change NOS | 3

ADVERSE EVENTS:
Time Frame: Adverse events collected on Days 1, 8 and 15 of each 21-day cycle and up to 30 days post-treatment.
Description: Patients were permitted to continue treatment in the absence of disease progression or intolerable toxicity. 25 patients received a median of 2 cycles (6 weeks) of treatment
Arm/Group | AUY922
Serious Adverse Events (participants affected / at risk) | 8/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AUY922 (N=25)
Gastrointestinal hemmorhage (Gastrointestinal disorders) | 3 (4)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Haemorrhage (Vascular disorders) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Feeding tube complication (Injury, poisoning and procedural complications) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AUY922 (N=25)
Abdominal pain (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 11
Diarrhea (Gastrointestinal disorders) | 16
Vomiting (Gastrointestinal disorders) | 7
Fatigue (General disorders) | 13
Alkaline phosphatase increased (Investigations) | 2
Asthenia (Musculoskeletal and connective tissue disorders) | 5
Blurred vision (Eye disorders) | 9
Flashing lights (Eye disorders) | 7
Delayed light/dark adaptation (Eye disorders) | 4
Decreased color perception (Eye disorders) | 2
Headache (Nervous system disorders) | 3
Anemia (Blood and lymphatic system disorders) | 10
Pain (Nervous system disorders) | 3
Anorexia (Gastrointestinal disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 2
Dysgeusia (Nervous system disorders) | 2
Night blindness (Eye disorders) | 3
Floaters (Eye disorders) | 2
Light sensitivity (Eye disorders) | 4
vision change NOS (Eye disorders) | 3 — NOS=not otherwise specified
Vision darkening (Eye disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.